CLINICAL TRIAL: NCT05375188
Title: To Evaluate if Dexmedetomidine Infusion Has a Role in Renal Protection in Patients Undergoing Coronary Artery Bypass Graft Surgery. A Randomized Control Trial
Brief Title: To Evaluate if Dexmedetomidine Infusion Provides Renal Protection in Patients Undergoing Coronary Artery Bypass Graft
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Institute of Cardiovascular Diseases, Pakistan (Other)
Responsible Party: Principal Investigator, Haris Tariq, Post Fellow, National Institute of Cardiovascular Diseases, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ERC- 66/2021
Record Dates: First submitted 2022-04-30; First posted 2022-05-16 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Dexmedetomidine; Hypnotics and Sedatives; Saline Solution

STUDY DESIGN:
Intervention Model Description: This study was conducted among 60 patients allocated randomly into two groups. In the study group (group D), dexmedetomidine was given as an infusion of 0.4 μg/kg/h from induction of anesthesia for 24 hours. In the control group (group C), the patients were receiving an equal volume of normal saline. The primary outcome of the study was Serum Creatinine (mg/dl) which was measured before the surgery as baseline and then at 48 hours after surgery.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group D (Experimental): Dexmedetomidine was given as an infusion of 0.4 μg/kg/h from induction of anesthesia for 24 hours.
  Interventions: Drug: Dexmedetomidine
- Group C (Placebo Comparator): Equal volume of normal saline.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Dexmedetomidine — DOSAGE FORM: IV Infusion DOSAGE: 0.4 mcg/kg/hr
  Other Names: sedatives (Precedex)
  Arms: Group D
Drug: Normal Saline — DOSAGE FORM: IV Infusion DOSAGE: Equal Volume
  Other Names: crystalloid fluid
  Arms: Group C

SUMMARY:
OBJECTIVE: Aim of this study is to follow and compare the changes in serum creatinine and urine output up to 48 hours of surgery in patients receiving dexmedetomidine infusion in addition to standard protocol (Experimental Group) as compared to the patients receiving standard protocol alone. (Control Group) in patients undergoing isolated coronary artery bypass grafting surgery (CABG) at a tertiary care cardiac center of Karachi, Pakistan.

STUDY DESIGN: Randomized control trial

PLACE & DURATION OF STUDY: The research will be conducted in the Department of Anesthesia & Intensive Care, National Institute of Cardiovascular Diseases (NICVD), Karachi. 6 months (01/08/2021 to 31/1/2022).

DATA COLLECTION PROCEDURE: This study was conducted among 60 patients allocated randomly into two groups. In the study group (group D), dexmedetomidine was given as an infusion of 0.4 μg/kg/h from induction of anesthesia for 24 hours. In the control group (group C), the patients were receiving an equal volume of normal saline.

PRIMARY OUTCOME: The primary outcome of the study was Serum Creatinine (mg/dl) which was measured before the surgery at baseline and then 48 hours after surgery.

SECONDARY OUTCOMES: The secondary outcomes were incidence of urine output per hour for up to 48 hours after surgery, operative time from induction of anesthesia till skin closure, aortic cross-clamp time from application of aortic cross-clamping till aortic declamping, CPB time from connecting the patient to extracorporeal circulation till termination of CPB, duration of ICU stay from transferring the patient from the operating room to the ICU till patient discharge to the ward, episodes of bradycardia and hypotension, dosage of inotropics and hemoglobin levels at baseline and up to 48 hours.

KEYWORDS: cardiac surgery-associated acute kidney injury, dexmedetomidine, serum creatinine.

DETAILED DESCRIPTION:
INTRODUCTION:

The incidence of cardiac surgery-associated acute kidney injury (CSA-AKI) varies from 5 to 42%.1 This percentage was found to be 7.86% according to study conducted in Pakistan. 2 Severe CSA-AKI is independently associated with three to eight-fold higher perioperative mortality, prolonged ICU and hospital length of stay, and increased cost of care.3 The etiology of renal injury is mainly due to elevation of renin levels as a result of sympathetic overactivity in addition to nephrotoxic inflammatory and hemodynamic components.4 The risk risk factors, even for those patients with complete renal recovery.3 As yet, there is no definite strategy for preventing AKI after cardiac surgery.5

Dexmedetomidine is a selective and potent α2-adrenoceptor agonist that is used for its anxiolytic, sedative, and analgesic properties.6 It decreases central nervous system sympathetic outflow in a dose-dependent manner and has opioid-sparing analgesic effects. There is increasing evidence of its organ-protective properties against ischemic and hypoxic injury, including cardioprotection, neuroprotection, and renoprotection.7,8 Peng et al. in his meta-analysis has highlighted the significant role of dexmedetomidine in reducing AKI after bypass surgeries.8 Then, R.Shi and H-T. Toe have also pointed out the promising renoprotective role of Dexmedetomidine in CABG surgeries. 10 Kidney Disease Improving Global Outcomes (KDIGO) is one of the latest classifications of identifying AKI and is commonly used in various studies. 11 In 2016, Ammar AS et al. in their study documented the reno-protective role of peri-operative dexmedetomidine infusion in cardiac surgery.4 The aim of this study is to use infusion of dexmedetomidine for renal protection in cardiac surgeries.

PATIENTS AND METHODS:

The aim of this study was to compare the changes in serum creatinine and urine output up to 48 hours of surgery in patients receiving dexmedetomidine infusion in addition to standard protocol as compared to the patients receiving standard protocol alone, and see if dexmedetomidine infusion reduced the incidence of Acute Kidney Injury (AKI) in patients undergoing coronary artery bypass graft surgery (CABG) in a tertiary cardiac center of Karachi, Pakistan. This study, a randomized control trial, was conducted in the Department of Anesthesia & Intensive Care, National Institute of Cardiovascular Diseases (NICVD), Karachi, for a period of 6 months (01/08/2021 to 31/1/2022), after approval from the ethical review committee of NICVD, Karachi.

Sample size for the study was calculated using G*Power version 3.1.9.2 using method of sample size calculation for two-sided hypothesis testing of two independent mean. Taking mean and standard deviation of serum creatinine after 48 hours of CABG in Dexmedetomidine and control group reported by Ammar AS et al. [3], at 5% level of significance and 90% power of test, the minimum required sample size of n=6 patients in each group was calculated. Considering the design effect, a sample size of 30 patients in each group was decided. N = 60 = 30 (control) + 30 (treatment).

Patients aged between 18 and 65 years, undergoing isolated coronary artery bypass grafting, and having ASA physical status class IV were included in the study. All patients with preoperative renal impairment (elevated creatinine and blood urea nitrogen levels), on diuretic use, preexisting hepatic or pulmonary disease, peripheral vascular disease, previous cardiac surgery, emergency surgery, reopening surgeries, surgeries requiring a deep hypothermic circulatory arrest, preoperative use of inotropes or vasopressors, perioperative use of diuretics, perioperative episode of CPR, preoperative hemoglobin level less than 12 mg/dl, hematological disorders and with morbid obesity were excluded.

Preoperatively, careful assessment of the cardiovascular system and investigations for the exclusion criteria and routine investigations which included complete blood count, coagulation profile, liver, and renal function tests, blood grouping, chest radiography, ECG, and echocardiography was done. On the day of surgery in the Operation Theatre (OT), wide bore intravenous cannula(16G) was inserted. Midazolam (0.01-0.02 mg/kg) was given as premedication. Arterial cannulation was applied under local anesthesia in the radial artery. In the operative room, pulse oximeter (SpO2), a five-lead ECG, and invasive arterial blood pressure monitoring was applied. Doses of induction was adjusted according to the hemodynamics and myocardial function of the patient. Anesthesia was induced by propofol (1-5 mg/kg) in addition to nalbuphine (0.1-0.2 mg/kg) and atracurium (0.6 mg/kg). After preoxygenation for 3 min and finally, a suitable-sized endotracheal tube was inserted, and the patient was connected to IPPV. Anesthesia was maintained with an inhalational agent (isoflurane) (1-2%) in 100% oxygen with the intent to maintain the mean arterial blood pressure and heart rate within 20% of the baseline. Atracurium will be administered, at a dose of 0.1-0.2 mg/kg to maintain muscle relaxation throughout the procedure. We divided a total of 60 patients after informed and written consent, in to two groups using computer generated random allocation based on Bernoulli distribution with probability of success (allocation of treatment group) as 0.50. In Dexmedetomidine Group (Group D), patients received Dexmedetomidine infusion in addition to standard management protocol (0.4 μg/kg/h from induction of anesthesia till the end of surgery). Whereas, in Control Group (Group C) patients allocated to this group will receive standard management protocol alone. We have used Kidney Disease Improving Global Outcomes (KDIGO) protocol in order to evaluate incidence of acute kidney injury. This protocol defines acute kidney injury as increase in serum creatinine more than 0.3mg/dl within 48 hours OR urine volume of less than 0.5ml/kg/hr for 6 hours. 12 After induction of anesthesia, central venous line, urinary catheter, and temperature probe was inserted. Before skin incision additional nalbuphine was injected. Arterial blood gases, serum Na and K, hematocrit, and blood glucose was measured after induction of anesthesia, during CPB, after weaning from CPB and according to needs. Activated clotting time was measured at baseline, 3 min after heparin administration, during CPB, and finally after reversal of heparin with protamine sulfate. The primary outcome of the study was Serum Creatinine (mg/dl) which was measured before the surgery at baseline and then 48 hours after surgery. The secondary outcomes were incidence of urine output per hour for up to 48 hours after surgery, operative time from induction of anesthesia till skin closure, aortic cross-clamp time from application of aortic cross-clamping till aortic declamping, CPB time from connecting the patient to extracorporeal circulation till termination of CPB, duration of ICU stay from transferring the patient from the operating room to the ICU till patient discharge to the ward, episodes of bradycardia and hypotension, dosage of inotropics and hemoglobin levels at baseline and then up to 48 hours. . Hypotension was defined as decrease in systolic blood pressure < 90mmHg.12 Bradycardia was defined as heart rate less than 60 beats/min. 12 The staff involved in the clinical care and members of the study group obtaining the data were blinded to randomization for the period of data achievement and analysis. Group allocation was revealed after the final statistical analysis.

Data was analyzed using IBM SPSS version 21, data was summarized by computing descriptive statistics such as mean ± SD for continuous response variables (including serum creatinine (ng/dL), urine output, and creatinine clearance) and frequency (%) for categorical response variables. Treatment and control group was compared for baseline characteristics and outcomes by conducting Chi-square test (for categorical variables) and independent sample t-test (for continuous response variables). Relative risk (95% CI) of AKI and other adverse outcomes were computed for treatment groups. Two-sided p-value of ≤ 0.05 was taken as criteria for statistical significance.

ELIGIBILITY:
Inclusion Criteria:

Ages ranged between 18 and 65 years.

* Patients undergoing isolated coronary artery bypass grafting.
* Class II and III ASA physical status.

Exclusion Criteria:

* Patients with preoperative renal impairment (elevated creatinine and blood urea nitrogen levels) and diuretic use.

  * Preexisting hepatic or pulmonary disease, peripheral vascular disease, previous cardiac surgery, emergency surgery, reopening surgeries, surgeries requiring a deep hypothermic circulatory arrest.
  * Preoperative use of inotropes or vasopressors.
  * Perioperative use of diuretics.
  * Perioperative episode of CPR.
  * Diabetic patients.
  * Preoperative hemoglobin level less than 12 mg/dl.
  * Hematological disorders.
  * Morbidly obese patients.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Post CABG Acute Kidney Injury at 48 hours | up to 48 hours post operatively
  Serum Creatinine (milligram/decilitre) as Kidney Disease Improving Global Outcomes criteria

SECONDARY OUTCOMES:
Aortic Cross Clamp Time | within 2 hours
  From to Aortic Clamping to Aortic Declamping
CPB Time | within 4 hours
  CPB time from connecting the patient to extracorporeal circulation till termination of CPB.
Time of Surgery | within 8 hours
  Operative Time from time of induction till skin closure
ICU stay | up to 48 hours
  Duration of ICU stay
Amount of Urine | up to 48 hours
  Urine Output (ml/hr)

CONTACTS AND LOCATIONS:
Overall Officials: Haris T Chohan, Principal Investigator — NICVD Karachi
Locations (1):
- NICVD Karachi, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
Only unique hospital ID of patients will be shared